CLINICAL TRIAL: NCT01260701
Title: A Phase II Study of MK-2206 (NSC-749607) as Second Line Therapy for Advanced Gastric and Gastroesophageal Junction Cancer
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Advanced Gastric or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02619; NCI-2011-02619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); SWOG-S1005; S1005; CDR0000689602; S1005 (Other: SWOG); S1005 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-11

CONDITIONS: Adenocarcinoma of the Gastroesophageal Junction; Diffuse Gastric Adenocarcinoma; Gastric Intestinal Type Adenocarcinoma; Gastric Mixed Adenocarcinoma; Recurrent Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (CLOSED TO ACCRUAL 05/01/13) (Experimental): Patients receive Akt inhibitor MK2206 PO every other day on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206

SUMMARY:
This phase II clinical trial studies how well Akt inhibitor MK2206 works in treating patients with advanced gastric or gastroesophageal junction cancer. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall survival (OS) for patients with advanced gastric and gastroesophageal junction (GEJ) adenocarcinoma treated with MK-2206 (Akt inhibitor MK2206).

SECONDARY OBJECTIVES:

I. To estimate the progression free survival (PFS) in this patient population. II. To estimate the response rate (confirmed and unconfirmed complete response [CR] and partial response [PR] by Response Evaluation Criteria In Solid Tumors [RECIST] 1.1) in this patient population.

III. To assess the frequency and severity of toxicity associated with this regimen.

OUTLINE (CLOSED TO ACCRUAL 05/01/13):

Patients receive Akt inhibitor MK2206 orally (PO) every other day on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma of the stomach or gastroesophageal (GE) junction that has progressed after first-line treatment, or is recurrent within 6 months after receiving adjuvant therapy; patients must have had exactly one prior systemic treatment regimen; previous adjuvant (chemotherapy [chemo]) radiotherapy is permitted; prior chemotherapy given concurrently with radiation for radiosensitization is not considered one prior systemic regimen
* Patients must have measurable disease; computed tomography (CT) scans or magnetic resonance imaging (MRIs) used to assess measurable disease must have been completed within 28 days prior to registration; CT scans or MRIs used to assess non-measurable disease must have been completed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form (RECIST 1.1)
* Patients must not have known brain metastases
* Patients must not have received chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to registration
* Patient must not have received prior treatment with a phosphatidylinositol 3 (PI3), v-akt murine thymoma viral oncogene homolog 1 (AKT) or mechanistic target of rapamycin (Mtor) inhibitor for any reason
* All toxicities from prior therapy must have resolved to =< grade 1 (Common Terminology Criteria for Adverse Events [CTCAE] version 4.0) prior to registration
* Patients must not be receiving or planning to receive any other investigational agents
* Patients must be able to tolerate oral medications and must not have malabsorption or chronic diarrhea (CTCAE version 4.0 grade 2 or higher); administration through a feeding tube is not permitted
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) both =< 2.5 x IULN; patients with liver metastases must have AST and ALT =< 5 x IULN
* Patients must have adequate kidney function as evidenced by at least ONE of the following:

  * Serum creatinine (mg/dL) =< IULN obtained within 14 days prior to registration
  * Calculated creatinine clearance > 50 ml/min; the serum creatinine value used in the calculation must have been obtained within 14 days prior to registration
* Patients must have international normalized ratio (INR) =< 1.2 unless taking therapeutic doses of warfarin; this result must be obtained within 14 days prior to registration
* Patients must have fasting blood sugar =< 150 mg/dL within 28 days prior to registration
* Patients must have hemoglobin A1C < 7% within 28 days prior to registration
* Patients must have an electrocardiogram (ECG) within 28 days prior to registration; patients must have corrected QT interval (QTcF) (by Fridericia's calculation) < 450 msec (male) or < 470 msec (female)
* Patients must have a Zubrod performance status of 0-1
* Patient must not have any of the following: a history of congenital long QT syndrome; use of concomitant medications that could prolong the QTc interval; New York Heart Association class III or IV heart failure; history of myocardial infarction within 6 months prior to registration; uncontrolled dysrhythmias; poorly controlled angina; resting heart rate =< 50 bpm (bradycardia)
* Patients must not be receiving concurrent treatment with drugs that are strong inducers or inhibitors of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4); patients must be able to safely discontinue treatment with these agents for >= 2 weeks prior to beginning protocol therapy
* Patient must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible
* Patient must not be pregnant or nursing; women/men of reproductive potential must have agreed to use two forms of contraception for the duration of protocol treatment and for one month after discontinuation of MK-2206; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any time a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ramesh Ramanathan, Principal Investigator — SWOG Cancer Research Network
Locations (187):
- United States (186):
  - Providence Hospital, Mobile, Alabama
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - The University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - The University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - NEA Baptist Memorial Hospital, Jonesboro, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Memorial University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - OnCare Hawaii-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Oncare Hawaii Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Cadence Cancer Center at Delnor, Geneva, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cadence Cancer Center in Warrenville, Warrenville, Illinois
  - Franciscan St. Francis Health-Beech Grove, Beech Grove, Indiana
  - Franciscan Saint Francis Health-Indianapolis, Indianapolis, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Hutchinson Regional Medical Center, Hutchinson, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - The University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Kansas City Cancer Centers-Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Kansas City Cancer Center-Shawnee Mission, Shawnee Mission, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium CCOP, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Truman Medical Center, Kansas City, Missouri
  - Kansas City Cancer Center - South, Kansas City, Missouri
  - Kansas City Cancer Centers - North, Kansas City, Missouri
  - Kansas City Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Frontier Cancer Center and Blood Institute-Billings, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Winthrop University Hospital, Mineola, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Cancer Control Consortium CCOP, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - McLeod Regional Medical Center, Florence, South Carolina
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Baylor Saint Luke's Medical Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - Memorial Hospital Of Martinsville, Martinsville, Virginia
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - EvergreenHealth Medical Center, Kirkland, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Cooperative of Puget Sound Oncology Consortium, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Wenatchee Valley Hospital and Clinics, Wenatchee, Washington
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- BCCA-Vancouver Cancer Centre, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Ramanathan RK, McDonough SL, Kennecke HF, Iqbal S, Baranda JC, Seery TE, Lim HJ, Hezel AF, Vaccaro GM, Blanke CD. Phase 2 study of MK-2206, an allosteric inhibitor of AKT, as second-line therapy for advanced gastric and gastroesophageal junction cancer: A SWOG cooperative group trial (S1005). Cancer. 2015 Jul 1;121(13):2193-7. doi: 10.1002/cncr.29363. Epub 2015 Mar 30. PMID 25827820

RESULTS

PARTICIPANT FLOW:
Groups:
- MK-2206: Patients receive Akt inhibitor MK-2206 PO QD, every other day, for 28 days. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | MK-2206
Started | 75
Eligible | 71
Eligible and Began Protocol Therapy | 70
Completed | 0
Not Completed | 75
Not completed — Adverse Event | 9
Not completed — Withdrawal by Subject | 2
Not completed — Progression | 53
Not completed — Death | 2
Not completed — Not protocol specified | 3
Not completed — Under review | 1
Not completed — Ineligible | 4
Not completed — Did not begin protocol therapy | 1

BASELINE CHARACTERISTICS:
Population: Eligible patients who began protocol therapy.
Arm/Group | MK-2206
Number analyzed (Participants) | 70
Age, Continuous [Median (Full Range); unit: years] | 60 [30 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  White | 62
  Asian | 5
  Unknown | 3

OUTCOME MEASURES:

1. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is measured from date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and without report of progression are censored at date of last contact. Progression is one or more of the following: 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed (over baseline if no decrease during therapy), as well as an absolute increase of at least 0.5 cm; unequivocal progression of non-measurable disease in the opinion of the treating physician; appearance of any new lesion/site; death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: Up to 2 years
Population: Eligible patients who began protocol therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MK-2206
Number analyzed (Participants) | 70
months | 1.8 [1.7 to 1.8]

2. Primary Outcome: Overall Survival (OS)
Description: Overall survival is calculated from date of registration to date of death due to any cause. Patients last known to be alive are censored at date of last contact.
Time Frame: Up to 2 years
Population: Eligible patients who began protocol therapy.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MK-2206
Number analyzed (Participants) | 70
months | 5 [4 to 9]

3. Secondary Outcome: Response Rate (Complete and Partial, Confirmed and Unconfirmed)
Description: Complete response (CR) is complete disappearance of all target and non-target lesions, no new lesions, and no disease related symptoms. Any lymph nodes must have reduction in short axis to < 1.0 cm. Partial response (PR) is >= 30% decrease under baseline of the sum of appropriate diameters of all target measurable lesions, no unequivocal progression of non-measurable disease, and no new lesions. Confirmed CR is two or more statuses of CR a minimum of four weeks apart documented before progression or symptomatic deterioration. Confirmed PR is two or more statuses of PR or better a minimum of four weeks apart documented before progression or symptomatic deterioration, but not qualifying as CR. Unconfirmed CR is one status of CR documented before progression or symptomatic deterioration but not qualifying as CR or PR. Unconfirmed PR is one status of PR documented before progression or symptomatic deterioration but not qualifying as CR, PR or unconfirmed CR.
Time Frame: Up to 2 years
Population: Eligible patients who began protocol therapy and were assessed for response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MK-2206
Number analyzed (Participants) | 68
percentage of participants | 1.5 [0 to 7.9]

4. Secondary Outcome: Number of Patients With Grade 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Any CTCAE 4.0 event of Grade 3 (severe), Grade 4 (life threatening), or Grade 5 (fatal) which were possibly, probably or definitely related to protocol treatment are included.
Time Frame: Up to 2 years
Population: Eligible patients who received any treatment and were assessed for adverse events are included in this summary.
Measure: Number; unit: Participants
Arm/Group | MK-2206
Number analyzed (Participants) | 70
Participants
  Adult respiratory distress syndrome | 1
  Alanine aminotransferase increased | 1
  Alkaline phosphatase increased | 2
  Allergic reaction | 1
  Anemia | 3
  Anorexia | 3
  Aspartate aminotransferase increased | 1
  Blood and lymphatic system disorders - Other | 1
  Blood bilirubin increased | 1
  Cardiac arrest | 1
  Dehydration | 1
  Dyspnea | 1
  Fatigue | 4
  Gastric hemorrhage | 1
  Gastroesophageal reflux disease | 1
  Hyperglycemia | 2
  Hypokalemia | 1
  Hyponatremia | 2
  Hypoxia | 1
  Lung infection | 1
  Lymphocyte count decreased | 1
  Nausea | 1
  Non-cardiac chest pain | 1
  Pleural effusion | 2
  Pneumonitis | 1
  Pruritus | 1
  Rash acneiform | 2
  Rash maculo-papular | 2
  Respiratory failure | 1
  Sinus bradycardia | 1
  Sinus tachycardia | 1
  Stroke | 1
  Upper gastrointestinal hemorrhage | 1
  Vomiting | 2

ADVERSE EVENTS:
Time Frame: Up to 2 years
Description: Eligible patients who received any treatment and were assessed for adverse events are included in the adverse event summaries.
Arm/Group | MK-2206
Serious Adverse Events (participants affected / at risk) | 31/70
Other Adverse Events (participants affected / at risk) | 67/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MK-2206 (N=70)
Anemia (Blood and lymphatic system disorders) | 4
Cardiac arrest (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colonic obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Esophageal hemorrhage (Gastrointestinal disorders) | 1
Gastric hemorrhage (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Obstruction gastric (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 2
Peritoneal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Creatinine increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9
Stroke (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK-2206 (N=70)
Anemia (Blood and lymphatic system disorders) | 22
Sinus bradycardia (Cardiac disorders) | 4
Abdominal distension (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 27
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 7
Dysphagia (Gastrointestinal disorders) | 10
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 32
Vomiting (Gastrointestinal disorders) | 19
Edema limbs (General disorders) | 4
Fatigue (General disorders) | 48
Fever (General disorders) | 4
Pain (General disorders) | 6
Alanine aminotransferase increased (Investigations) | 8
Alkaline phosphatase increased (Investigations) | 21
Aspartate aminotransferase increased (Investigations) | 11
Blood bilirubin increased (Investigations) | 4
Creatinine increased (Investigations) | 7
Electrocardiogram QT corrected interval prolonged (Investigations) | 8
Lymphocyte count decreased (Investigations) | 14
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 18
White blood cell decreased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 27
Dehydration (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 28
Hypoalbuminemia (Metabolism and nutrition disorders) | 12
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypokalemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 9
Anxiety (Psychiatric disorders) | 8
Depression (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 13
Pruritus (Skin and subcutaneous tissue disorders) | 16
Rash acneiform (Skin and subcutaneous tissue disorders) | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less